CLINICAL TRIAL: NCT04547647
Title: Back Deformity Among Adolescent Students in Elkharga City- The New Vally Governorate- Egypt
Brief Title: Back Deformity in Adolescents Students
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dalia Mahran, Doctor, Assiut University
Other Study IDs: Back deformity in adolescents
Record Dates: First submitted 2019-09-30; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2019-09

CONDITIONS: Back Disorder
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: X- Ray — X-Ray with A-P and lateral view of the whole spine.

SUMMARY:
1. Determine the prevalence of scoliosis and kyphosis among male adolescents in preparatory and secondary governmental schools in El Kharga city.
2. To identify factors affecting aetiology and morphology of scoliosis and kyphosis among male adolescents in governmental preparatory and secondary schools in El Kharga city.
3. To assess the effect of scoliosis and kyphosis among male adolescents in governmental preparatory and secondary schools in El Kharga city on related life style aspects.

DETAILED DESCRIPTION:
The anterior and posterior curves of concavity are part of the physiological position of the spinal column, and are represented by cervical lordosis, thoracic kyphosis, lumbar lordosis, and new sacral and coccygeal kyphosis. Despite all these curves, the spinal column should work mechanically as a straight and rigid axis to withstand stress, and should be functionally flexible in order to allow movement. This mix of opposite behaviors (rigidness and flexibility) is the result of a complex stabilization system formed by muscles that contract and relax harmonically and absorb any impact exerted on the spinal column structure. Biomechanically speaking, the spinal column influences and is influenced by positioning and stress of the pelvic and scapular belts, and upper and lower limbs, respectively. Postural deformities and alterations should not be evaluated only in terms of bone structure, but also in terms of the functional assembly represented by the spinal column [2].

Adolescence is a stage of fast physical development in which the nervous system and musculoskeletal system have yet to fully develop. Changes in the physical morphology of the spine are known to cause musculoskeletal system conditions, such as non-specific back pain. Moreover, the spinal morphology as scoliosis and kyphosis.

With early identification and intervention, scoliosis may be prevented from progressing, so that it does not interfere with mobility, activity or comfort. Scoliosis has a large percentage that remains asymptomatic,[4] Therefore the feasibility of screening is worthwhile

ELIGIBILITY:
Inclusion Criteria:

* Male students from the 2nd and 3rd preparatory levels and 1st secondary level

Exclusion Criteria:

* female students

Ages: 14 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Male students from the 2nd and 3rd preparatory levels and 1st secondary level will be included.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | 3 month
  Self administrated questionnaire

REFERENCES:
- [Background] Theroux J, Stomski N, Hodgetts CJ, Ballard A, Khadra C, Le May S, Labelle H. Prevalence of low back pain in adolescents with idiopathic scoliosis: a systematic review. Chiropr Man Therap. 2017 Apr 20;25:10. doi: 10.1186/s12998-017-0143-1. eCollection 2017. PMID 28439404
- [Background] Feng Q, Jiang C, Zhou Y, Huang Y, Zhang M. Relationship between spinal morphology and function and adolescent non-specific back pain: A cross-sectional study. J Back Musculoskelet Rehabil. 2017;30(3):625-633. doi: 10.3233/BMR-160544. PMID 28234252